CLINICAL TRIAL: NCT06857721
Title: Evaluation of Intraoral Scanners in Terms of Comfort in Pediatric Patients: A Crossover Randomized Trial
Brief Title: Comfort Assessment of Intraoral Scanners in Children
Acronym: RCT-CS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batman University (Other)
Responsible Party: Principal Investigator, Nursezen Kavasoglu, Assistant Professor Dr., Batman University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NK01
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Intraoral Scanner

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital scanner group (Experimental): It consists of children whose digital measurements were taken with the Itero scanner in the first appointment and with the 3Shape scanner in the second appointment.
  Interventions: Device: Intraoral Scanners

INTERVENTIONS:
Device: Intraoral Scanners — Intraoral scanners for pediatric patients

SUMMARY:
With the advancement of the digital age, dentistry has been one of the fields that has benefited most from technological innovations. Among these advancements, digital intraoral scanners, which precisely capture the three-dimensional geometry of objects, have become widely used, particularly in prosthodontics and orthodontics. The increasing integration of digitalization in pediatric dentistry has also improved treatment processes, making them more efficient and comfortable for both patients and clinicians.

Previous studies comparing conventional and digital impression techniques suggest that patients generally prefer digital scanning due to improved comfort and reduced procedural time. However, research on pediatric patients remains limited, with most studies focusing on general performance rather than specific patient experiences. Given the unique anatomical and psychological characteristics of children, a comprehensive evaluation of comfort perception in different intraoral scanners is necessary.

This study aims to assess the effects of two different intraoral scanners on pediatric patients' comfort perception. It is designed as a single-center, randomized controlled crossover study, approved by the Ethics Committee of the Faculty of Dentistry at Batman University. A total of 68 children meeting the inclusion criteria were recruited and randomly assigned to undergo intraoral scanning with two different devices (IteroTM and 3ShapeTM) at separate visits. Comfort levels were assessed using the Animale Emoji Scale (AES), a validated tool for measuring children's emotional responses to procedures.

By comparing the comfort perception of different intraoral scanners in pediatric patients, this study aims to provide evidence-based guidance for clinicians in selecting the most patient-friendly digital impression techniques, ultimately improving patient experience and clinical workflow in pediatric dentistry.

To prevent bias during the procedure, the intraoral scan was performed using either the Itero™ or 3Shape™ device, determined by simple randomization. Since the sample consisted of consecutive cases, random selection was performed by coin toss.

At the first appointment, parents or legal guardians were informed about the study, a consent form was provided, and they were informed that they would be contacted again if they wished to participate. The first scan was performed using the Itero Element 2D (Align Technology, San Jose, CA, USA) device.

The second appointment was scheduled 7 to 30 days after the initial appointment to avoid affecting children's comfort, in accordance with previous studies. The second scan was planned using the 3Shape Trios 3 (3Shape, Copenhagen, Denmark) device.

All intraoral scans were performed by the principal investigator of the study. According to the manufacturer's instructions, the patient was scanned in a supine position following the same sequence (lower jaw, upper jaw, and bite registration).

To increase the reliability of the results, all measurements were taken by a single experienced researcher who took at least 100 measurements with both scanning devices. To ensure standardization, all patients were positioned at 11 o'clock relative to the unit and the scanning device was positioned at 1 o'clock for all scans.

The primary outcome of the study was patient comfort. Participants' comfort was measured using the Animated Emoji Scale (AES) based on questions prepared during the procedure. Children were asked to select the face that best reflected their feelings after the procedure (Figure 1). For younger children, the AES scale was completed under the supervision of the operator and with guiding questions. The AES scale includes 6 different facial expressions ranging from "no pain" to "worst pain," and each face is scored from 0-2-4-6-8-10. These measurements were always taken by the same observer.

Sample size was calculated using G*Power, and data analysis was performed using IBM SPSS 21® Software (Armonk, NY, USA). The normality of the data was evaluated using the Shapiro-Wilk's and/or Kolmogorov Smirnov tests. The significance level was set at p<0.05. In case of deviation from the normal distribution, differences between groups were examined using the Mann Whitney U and Kruskal Wallis-H tests. In case of a significant difference in the Kruskal Wallis-H test, a Post-Hoc multiple comparison test was applied. Differences between two dependent variables were analyzed using the Wilcoxon test.

ELIGIBILITY:
Inclusion Criteria:

Healthy children Children have no experience with dental measurement techniques or intraoral scanning.

Exclusion Criteria:

Children with craniofacial syndromes Children with systemic diseases Children with Behavioral problems

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Differences Between Genders in Children's Responses During Measurements Made with the IteroTM | 15 minutes

SECONDARY OUTCOMES:
Differences Between Genders in Children's Responses During Measurements Made with the 3ShapeTM | 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Dental In Oral and Dental Health Polyclinic, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol
Time Frame: Start Date: 04.2025 End Date: 07.2025
Access Criteria: Dentists